CLINICAL TRIAL: NCT05571475
Title: The Effect of Simulated Competition on Repeated-sprint Cycling Performance and on Measures of Physiological and Psychological Stress.
Brief Title: The Effects of Simulated Competition on Repeated-sprint Cycling Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: StMarysUC6
Record Dates: First submitted 2022-09-07; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulated competition (Experimental): During the experimental condition, the participants will be competing for a reward, will be given verbal encouragement, and will receive performance feedback.
  Interventions: Other: Simulated competition
- Control (No Intervention): During the control condition, the participants will be asked to sprint without verbal encouragement or any performance feedback.

INTERVENTIONS:
Other: Simulated competition — During a competition, athletes will typically compete for a reward, against opponents and in the presence of others. This will be replicated in the laboratory.
  Arms: Simulated competition

SUMMARY:
Sprint cycling performance has been found to be reduced when two sprints were undertaken 12 minutes apart. In a follow-up study, the investigators found evidence to suggest that some of the loss in performance that was experienced in the second sprint was due to a psychological, rather than a physiological, limitation. It is conceivable that this loss in performance would not exist during a competition. The aim of this study is, therefore, to investigate the influence that a competitive environment has on repeated-sprint performance.

ELIGIBILITY:
Inclusion Criteria:

* regular strength/sprint training (at least 2 sessions per week)

Exclusion Criteria:

* Injured or a contraindicative medical condition

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Sprint Power Output | From baseline to completion, ~42 days
  The Lode Excalibur Sport cycle ergometer records power output at 5Hz. Peak power output will be defined as the highest power output recorded. Mean power output will be calculated as the average power output over the 27 s sprint. Comparisons will be made between conditions.

SECONDARY OUTCOMES:
Heart-rate Variability | From baseline to completion, ~42 days
  Heart-rate variability provides a measure of physiological stress. Recordings will be taken at rest, after the warm-up, and following the sprints. Comparisons will be made between conditions.
Salivary Concentration of Alpha Amylase | From baseline to completion, ~42 days
  Alpha amylase is a digestive enzyme found in saliva. Alpha amylase also provides a measure of physiological stress. Recordings will be taken at rest, after the warm-up, and following the sprints. Comparisons will be made between conditions.
20 cm Visual Analogue Scale to Assess Anxiety | From baseline to completion, ~42 days
  The scale will range from not at all anxious to very anxious. Participants will be asked to indicate how anxious they feel by place a clear mark on the scale. Measurements will be taken at rest, after the warm-up, and following the sprints. Comparisons will be made between conditions.
20 cm Visual Analogue Scale to Assess Self-efficacy | From baseline to completion, ~42 days
  The scale will range from cannot do it at all to highly certain. Participants will be asked about their confidence in their ability to improve on their baseline sprint performance. Measurements will be taken just prior to each sprint. Comparison to baseline.
Sport Anxiety Scale-2 - a questionnaire to assess cognitive and somatic anxiety. | Baseline
  Measured once. Correlation will performance. The response for each question carries a score of between 1 and 4. A higher number is reflective of a greater level of anxiety.